CLINICAL TRIAL: NCT02676479
Title: The Histological and Genetic Investigation of Cells, Fluid and Tissue in the Uterine Cavity, Using the Uterine Irrigation Method, in Patients Who Suffer From Unexplained Infertility and Hereditary Genetic Disease, and Who Require PGD Scans.
Brief Title: Uterine Irrigation Method in Infertility Patients Who Require PGD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University (Other)
Collaborators: Previvo Genetics (Industry); Acibadem Fulya Hospital (Other)
Responsible Party: Principal Investigator, Ercan Bastu, Associate Professor of Obstetrics and Gynecology, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016
Record Dates: First submitted 2016-01-23; First posted 2016-02-08 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pre-Implantation Embryo Recovery; Genetic Diseases, Inborn
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uterine Lavage Group (Experimental): The study will involve up to 30 pairs of male and female sexually intimate partners who are carriers for a genetic disease (e.g Sickle Cell Disease or Thalassemia) and at high risk of transmitting the gene.
  The female partner will be superovulated to mature multiple oocytes which can be fertilized, inseminated with her partner's sperm through intra-uterine insemination (IUI). Four to six days after IUI, the female partner will undergo a non-surgical uterine lavage procedure (Previvo Uterine Lavage System™, CA, U.S.A.) to recover preimplantation embryos.
  Interventions: Device: Uterine Lavage Group

INTERVENTIONS:
Device: Uterine Lavage Group — The PI places the Lavage Catheter per instructions for use
  * Use of a tenaculum or cervical stitch is required
  * Use of saline to wash the cervix is required
  * Use of abdominal ultrasound guidance with a full bladder is required The PI records if there was clinically significant fluid loss through the cervix.

SUMMARY:
The study will involve up to 30 pairs of male and female sexually intimate partners who are carriers for a genetic disease (e.g Sickle Cell Disease or Thalassemia) and at high risk of transmitting the gene. The female partner will be superovulated to mature multiple oocytes which can be fertilized, inseminated with her partner's sperm through intra-uterine insemination (IUI). Four to six days after IUI, the female partner will undergo a non-surgical uterine lavage procedure to recover preimplantation embryos.

DETAILED DESCRIPTION:
The study is a prospective, single center, single-arm study to evaluate healthy cells which do not carry illnesses, by collecting and performing the histological and genetic analyses of blastocysts, endometrial tissue and cells, which have been formed in the uterus, without any burden of the morbidity and mortality caused by the oocyte collection process, and which thereby have not been subjected to any iatrogenic intervention, with uterine lavage.

The study will involve up to 30 pairs of male and female sexually intimate partners who are carriers for a genetic disease (e.g Sickle Cell Disease or Thalassemia) and at high risk of transmitting the gene.

The female partner will be superovulated to mature multiple oocytes which can be fertilized, inseminated with her partner's sperm through intra-uterine insemination (IUI). Four to six days after IUI, the female partner will undergo a non-surgical uterine lavage procedure to recover preimplantation embryos.

Following lavage, a GnRH antagonist will be administered to cause lysis of multiple corpora lutea to mitigate risk of hyperstimulation from the use of fertility medication and reduce the risk of ectopic pregnancy should the lavage procedure not recover all preimplantation embryos.

Recovered preimplantation embryos may be screened for aneuploidy and genetic disease, then cryopreserved for potential future use by the subjects and the Investigator separate from the purpose of this study.

Each subject participates in the trial for up to 10-20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Female Age 21-39 years old.
* BMI between 18-35 kg/m2
* Presence of a normal uterine cavity, both fallopian tubes and their respective ovaries as assessed by hysterosalpingogram and/or sonohysterogram (SHG).
* Regular menstrual cycles every 26-32 days
* Male partner aged 21-40 yrs with a normal semen analysis.
* Infertile couples, which carry hereditary genetic diseases and genetic anomalies, and have a high probability of passing these on to their children.

Exclusion Criteria:

* Any active, uncontrolled, clinically significant medical condition as determined by the treating principal investigator
* Previous history of prior appendectomy and/or lower abdominal surgery
* Previous history of prior tubal surgery or ectopic pregnancy
* Contraindication for the use of oral contraceptive pills
* Clinically significant abnormal basic metabolic panel lab results
* Positive test or history of any of the following conditions:
* Human immunodeficiency virus (HIV)
* Hepatitis B infection
* Hepatitis C infection
* Syphilis (RPR)
* Chlamydial pelvic infection
* Gonorrheal pelvic infection.
* Positive Pregnancy Test
* No prior IUD for 60 days and not currently in place

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blastocyst Retrieval | 3 months
  Number of blastocyst retrieved

SECONDARY OUTCOMES:
Blastocyst Quality | 3 months
  Number of cells developed in each blastocyst

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bastu, MD,AssocProf, Principal Investigator — Istanbul University School of Medicine
Locations (1):
- Istanbul University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/4037016